CLINICAL TRIAL: NCT03706183
Title: The Evaluation of the Ischemia-modified Albumin Levels in the Patients With Sudden Sensorineural Hearing Loss
Brief Title: Ischemia- Modified Albumin Levels in the Sudden Hearing Loss
Acronym: IMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ufuk Düzenli, Principal Investigator, Assistant Professor, Yuzuncu Yil University
Other Study IDs: YYU7139
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Sudden Hearing Loss; Ischemia
MeSH Terms: conditions — Hearing Loss, Sudden; Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group: The IMA levels will be determined and the association of the IMA and Hearing thresholds will be evaluated.
  Interventions: Diagnostic Test: Ischemia-modified albumin; Diagnostic Test: Hearing thresholds
- Control Group: The IMA levels will be determined.
  Interventions: Diagnostic Test: Ischemia-modified albumin; Diagnostic Test: Hearing thresholds

INTERVENTIONS:
Diagnostic Test: Ischemia-modified albumin — The biomarker was investigated in many studies and it was associated with the ischemia and tissue injury.
Diagnostic Test: Hearing thresholds — The hearing levels will be determined for each group.
  Other Names: audiologic assessment

SUMMARY:
To evaluate ischemia-modified albumin levels in these patients to investigate the presence of ischemia in patients presenting with sudden hearing loss.

DETAILED DESCRIPTION:
Sudden hearing loss is an ENT emergence occurring within 72 hours, with sensorineural hearing loss of more than 30 dB on three consecutive frequencies. The incidence of this disease was 5-20 / 100000. The etiology of this disease has not been fully elucidated. In addition, viral infections, tumors, autoimmune diseases and vascular insufficiency have been suggested as etiologic factors by different researchers. There is no definitive routine treatment modality in the world because the etiology is not fully established. However, corticosteroid treatment is a well-accepted agent for the treatment of internal ear damage. In recent years, studies have shown that ischemia has an important place in etiology and hyperbaric oxygen therapy has become one of the routine treatment protocols. Another important point in terms of the prognosis of the disease is that spontaneous recovery of sudden hearing loss in 30-70% of the patients is observed in different studies.

Ischemia-modified albumin is a compound used as a marker of oxidative stress and used to determine the severity of cardiac ischemia.

In this study, the levels of ischemia-modified albumin levels in patients with SSHL and healthy control patients will be measured and their effectiveness in revealing the etiology of SSHL will be investigated. The difference between ischemia-modified albumin between patients and healthy control subjects will be evaluated. The number of patients and control groups shall be 30 individuals.

The evaluation of the hearing of the patients with hearing loss will be performed by the Otorhinolaryngology Department of Yuzuncu Yıl University. The study is planned to be performed with a total of 30 patients aged 18-50 years. Those who are diagnosed with SSHL will be included in the group and chronic diseases in the ear will be excluded. Thirty healthy patients with similar age and gender will be included in the study as the control group. The patients in the control group, must have normal hearing levels. The amounts of ischemic modified albumin in the study group and in the control group will be measured. Hearing levels will be determined at the admission time and 3,7,10th days and 1st month. 5 ml of peripheral blood samples taken from both groups of patients will be taken into biochemistry tubes. The blood will be centrifuged at 4000 rpm for 5 minutes to separate from the serum and plasma. Serum samples obtained will be stored at -20 oC until analysis. The selected samples are not hemolyzed and lipemic. Once the target number has been reached, all samples will be carefully mixed and then returned to the room temperature (15ına18 oC). It will be examined on the same day to avoid any differences between all sera. Statistical analysis will be done and interpreted.

ELIGIBILITY:
Inclusion Criteria:

* Admission with sensorineural hearing loss

Exclusion Criteria:

* cardiovascular disease
* hypertension
* diabetes mellitus
* malignancy
* chronic inflammatory disease
* kidney failure
* liver failure

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study group will include the patients with SSHL and control group will include the healthy controls with normal hearing thresholds
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
ischemia-modified albumin levels | 1 month
  The investigators will measure the levels of the IMA in the patients with SSHL and control group participants. The measurements will be done at the 1,3, 7 and 10th days and 1st month after diagnosing the SSHL. One measurement will be performed for the control group participants.
hearing thresholds | 1 month
  The hearing levels will be determined by an audiologist. The hearing determinations will be performed at the day when IMA measurements will be done for each group.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim JH, Roh KJ, Suh SH, Lee KY. Improvement of sudden bilateral hearing loss after vertebral artery stenting. J Neurointerv Surg. 2016 Mar;8(3):e12. doi: 10.1136/neurintsurg-2014-011595.rep. Epub 2015 Feb 24. PMID 25712982
- [Result] Onal M, Elsurer C, Selimoglu N, Yilmaz M, Erdogan E, Bengi Celik J, Kal O, Onal O. Ozone Prevents Cochlear Damage From Ischemia-Reperfusion Injury in Guinea Pigs. Artif Organs. 2017 Aug;41(8):744-752. doi: 10.1111/aor.12863. Epub 2017 Mar 5. PMID 28261890
- [Result] Kilic MO, Guldogan CE, Balamir I, Tez M. Ischemia-modified albumin as a predictor of the severity of acute appendicitis. Am J Emerg Med. 2017 Jan;35(1):92-95. doi: 10.1016/j.ajem.2016.10.010. Epub 2016 Oct 7. PMID 27769665
- [Result] Can S, Akdur O, Yildirim A, Adam G, Cakir DU, Karaman HI. Myelin basic protein and ischemia modified albumin levels in acute ischemic stroke cases. Pak J Med Sci. 2015 Sep-Oct;31(5):1110-4. doi: 10.12669/pjms.315.7702. PMID 26648996